CLINICAL TRIAL: NCT00783718
Title: A Phase 3, Randomized, Placebo-Controlled, Blinded, Multicenter Study of the Induction and Maintenance of Clinical Response and Remission by MLN0002 in Patients With Moderate to Severe Ulcerative Colitis
Brief Title: Study of Vedolizumab (MLN0002) in Patients With Moderate to Severe Ulcerative Colitis
Acronym: GEMINI I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C13006; U1111-1156-8422 (Registry Identifier: WHO); 2008-002782-32 (EudraCT Number); NL25207.096.08 (Registry Identifier: CCMO); CTRI/2009/091/000128 (Registry Identifier: CTRI); NMRR-08-1046-2201 (Registry Identifier: NMRR); C13006CTIL (Other: Israel MoH); 09/H1102/66 (Registry Identifier: NRES)
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab; LDP-02

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vedolizumab (Experimental): In the Induction Phase participants received vedolizumab 300 mg, administered by intravenous infusion at Week 0 and Week 2 (Days 1 and 15).
  In the Maintenance Phase, participants who demonstrated a clinical response at Week 6 according to protocol-specified criteria were randomized in a 1:1:1 ratio to double-blind treatment with vedolizumab administered every 4 weeks, vedolizumab administered every 8 weeks, or placebo for up to Week 50. Participants who did not demonstrate response at Week 6 of the Induction Phase continued treatment with vedolizumab, administered every 4 weeks during the Maintenance Phase.
  Interventions: Drug: vedolizumab
- Placebo (Placebo Comparator): In the Induction Phase participants received placebo intravenous infusion at Week 0 and Week 2 (Days 1 and 15). Participants continued to receive placebo during the Maintenance Phase, regardless of treatment response during Induction.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: vedolizumab — Vedolizumab for intravenous infusion
  Other Names: Entyvio; MLN0002; MLN02; LDP-02
  Arms: Vedolizumab
Other: Placebo — Placebo intravenous infusion
  Arms: Placebo

SUMMARY:
The primary purpose of this study was to determine the effect of vedolizumab induction treatment on clinical response at 6 weeks and to determine the effect of vedolizumab maintenance treatment on clinical remission at 52 weeks.

DETAILED DESCRIPTION:
This multicenter, phase 3, randomized, blinded, placebo-controlled study in patients with moderately to severely active ulcerative colitis comprises two phases:

* The Induction Phase, designed to establish the efficacy and safety of vedolizumab for the induction of clinical response and remission.
* The Maintenance Phase, designed to establish the efficacy and safety of vedolizumab for the maintenance of clinical response and remission.

The 6-week Induction Phase contained 2 cohorts of participants: Cohort 1 participants were randomized and treated with double-blind study drug, and Cohort 2 participants were treated with open-label vedolizumab. The second cohort was enrolled to ensure that the sample size of Induction Phase responders randomized into the Maintenance Study provided sufficient power for the Maintenance Study primary efficacy analysis. These participants did not contribute to the efficacy analyses performed for the Induction Study. Participants in both cohorts were assessed for treatment response at Week 6.

In the Maintenance Phase vedolizumab-treated participants from both Cohort 1 and Cohort 2 who demonstrated a clinical response were randomized in a 1:1:1 ratio to double-blind treatment with vedolizumab administered every 4 weeks (Q4W), vedolizumab administered every 8 weeks (Q8W), or placebo. Vedolizumab-treated participants who did not demonstrate response at Week 6 continued treatment with open-label vedolizumab, administered Q4W. Participants treated with double-blind placebo in the Induction Phase continued on double-blind placebo during the Maintenance Phase, regardless of treatment response during induction. The Maintenance Phase began at Week 6 and concluded with Week 52 assessments.

After the Week 52 assessments, participants meeting protocol-defined criteria were eligible to enroll in Study C13008 (NCT00790933; Long-term Safety) to receive open-label vedolizumab treatment. Participants who withdrew early (prior to Week 52) due to sustained nonresponse, disease worsening, or the need for rescue medications may also have been eligible for Study C13008. Participants who did not enroll into Study C13008 were to complete a final on-study safety assessment at Week 66 (or final safety visit 16 weeks after the last dose) in the Maintenance Phase of Study C13006.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

1. Diagnosis of moderately to severely active ulcerative colitis
2. Demonstrated, over the previous 5 year period, an inadequate response to, loss of response to, or intolerance at least 1 of the following agents:

   1. Immunomodulators
   2. Tumor necrosis factor-alpha (TNFα) antagonists
   3. Corticosteroids
3. May be receiving a therapeutic dose of conventional therapies for inflammatory bowel disease (IBD) as defined by the protocol

Exclusion Criteria:

1. Evidence of abdominal abscess at the initial screening visit
2. Extensive colonic resection, subtotal or total colectomy
3. Ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine
4. Have received non permitted IBD therapies within either 30 or 60 days, depending on the medication, as stated in the protocol
5. Chronic hepatitis B or C infection
6. Active or latent tuberculosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 895 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (105):
- United States (102):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Apex Clinical Trials, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Gastrointestinal Bioscience, Los Angeles, California
  - Paramount Medical Specialty, Montebello, California
  - Capital Gastroenterology Consultants Medical Group, Sacramento, California
  - Clinical Applications Laboratories Inc., San Diego, California
  - Desta Digestive Disease Medical Center, San Diego, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Gastroenterology of the Rockies, Lafayette, Colorado
  - Rocky Mountain Gastroenterology Associates P.L.L.C., Lakewood, Colorado
  - Arapahoe Gastroenterology Associates P.C, Littleton, Colorado
  - South Denver Gastroenterology, Lone Tree, Colorado
  - Lynn Institute of Pueblo, Pueblo, Colorado
  - Gastroenterology Center of Connecticut, P.C., Hamden, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Florida, Jacksonville, Jacksonville, Florida
  - East Coast Institute for Research, Jacksonville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Osler Clinical Research, Melbourne, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - United Medical Research Institute, New Smyrna Beach, Florida
  - Compass Research LLC, Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - West Wind'r Research & Development, LLC, Tampa, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Southeast Regional Research Group, Columbus, Georgia
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Digestive Research Associates, Newnan, Georgia
  - St. Joseph's/Candler Health System, Savannah, Georgia
  - DLW Research System, Snellville, Georgia
  - Carle Clinic Association P.C., Urbana, Illinois
  - Digestive & Liver Consultants, Clive, Iowa
  - Iowa Digestive Disease Center, Clive, Iowa
  - University Of Kansas, Kansas City, Kansas
  - Cotton O'Neil Digestive Health Center, Topeka, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University Of Louisville, Louisville, Kentucky
  - Gastroenterology Associates, Baton Rouge, Louisiana
  - University of Maryland Medical Group, Baltimore, Maryland
  - Metropolitan Gastroenterology Group, P.C., Chevy Chase, Maryland
  - Shah Associates, Prince Frederick, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - The Center for Clinical Studies, Dearborn, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Gastroenterology Associates of Western Michigan, P.L.C., Wyoming, Michigan
  - Minnesota Gastroenterology, P.A., Plymouth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Truman Medical Center, Kansas City, Missouri
  - Center for Digestive and Liver Diseases, Inc., Mexico, Missouri
  - Washington University, St Louis, Missouri
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Affiliates in Gastroenterology PA, Morristown, New Jersey
  - University of Medicine and Dentistry of New Jersey-NJMS, New Brunswick, New Jersey
  - The Gastroenterology Group of South Jersey, Vineland, New Jersey
  - Hepatobiliary Associates of New York, Bayside, New York
  - Digestive Health Physician, Cheektowaga, New York
  - Long Island Clinical Research Associates, Great Neck, New York
  - Long Island Gastroenterology Group, P.C., Merrick, New York
  - New York Presbyterian Hospital, New York, New York
  - Present Chapman Marion Steinlauf MD PC, New York, New York
  - Kim, Chung MD (Private Practice), Pittsford, New York
  - University of Rochester, Rochester, New York
  - Long Island Digestive Disease Consultants, Setauket, New York
  - SUNY Stony Brook University Medical Center, Stony Brook, New York
  - Syracuse Gastroenterological Associates, Syracuse, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Charlotte Gastroentology and Hepatology, P.L.L.C, Charlotte, North Carolina
  - Northwest Piedmont Clinical Research, Inc., Elkin, North Carolina
  - Burke Research Associates, Morganton, North Carolina
  - Consultants for Clinical Research Inc., Cincinnati, Ohio
  - Dayton Science Institute, Dayton, Ohio
  - Options Health Research, Tulsa, Oklahoma
  - The Oregon Clinic-West Hills Gastroenterology, Portland, Oregon
  - University of Pittsburgh Medical Center - Cancer Centers, Pittsburgh, Pennsylvania
  - Medical University Of SC CAR, Charleston, South Carolina
  - Gastroenterology Center of the MidSouth, PC, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Austin Gastroenterology, PA, Austin, Texas
  - Bayou City Research, Ltd., Houston, Texas
  - Baylor College Of Medicine, Houston, Texas
  - Gastroenterology Consultants, Houston, Texas
  - Jacon Medical Research Associates, Houston, Texas
  - Digestive Health Center, Pasadena, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Gastroenterology Clinic of San Antonio, San Antonio, Texas
  - Stone Oak Research Foundation, San Antonio, Texas
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - Granite Peaks Gastroenterology, Sandy City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Gastroenterology Associates of Northern Virginia, Fairfax, Virginia
  - Digestive and Liver Disease Specialist Ltd, Norfolk, Virginia
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Puget Sound Medical Research, Edmonds, Washington
  - Pharmaseek, LLC, Madison, Wisconsin
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Zeidler Ledcor Center-Univerisity of Alberta, Edmonton, Alberta
  - Royal University Hospital, Saskatoon, Saskatchewan
- Pharmaseek, LLC, Ponce, Puerto Rico

REFERENCES:
- [Result] Feagan BG, Rutgeerts P, Sands BE, Hanauer S, Colombel JF, Sandborn WJ, Van Assche G, Axler J, Kim HJ, Danese S, Fox I, Milch C, Sankoh S, Wyant T, Xu J, Parikh A; GEMINI 1 Study Group. Vedolizumab as induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2013 Aug 22;369(8):699-710. doi: 10.1056/NEJMoa1215734. PMID 23964932
- [Derived] Dulai PS, Feagan BG, Sands BE, Chen J, Lasch K, Lirio RA. Prognostic Value of Fecal Calprotectin to Inform Treat-to-Target Monitoring in Ulcerative Colitis. Clin Gastroenterol Hepatol. 2023 Feb;21(2):456-466.e7. doi: 10.1016/j.cgh.2022.07.027. Epub 2022 Aug 4. PMID 35934286
- [Derived] Wyant T, Yang L, Rosario M. Comparison of the ELISA and ECL Assay for Vedolizumab Anti-drug Antibodies: Assessing the Impact on Pharmacokinetics and Safety Outcomes of the Phase 3 GEMINI Trials. AAPS J. 2020 Nov 16;23(1):3. doi: 10.1208/s12248-020-00518-0. PMID 33200296
- [Derived] Okamoto H, Dirks NL, Rosario M, Hori T, Hibi T. Population pharmacokinetics of vedolizumab in Asian and non-Asian patients with ulcerative colitis and Crohn's disease. Intest Res. 2021 Jan;19(1):95-105. doi: 10.5217/ir.2019.09167. Epub 2020 Jul 10. PMID 32635680
- [Derived] Loftus EV Jr, Sands BE, Colombel JF, Dotan I, Khalid JM, Tudor D, Geransar P. Sustained Corticosteroid-Free Clinical Remission During Vedolizumab Maintenance Therapy in Patients with Ulcerative Colitis on Stable Concomitant Corticosteroids During Induction Therapy: A Post Hoc Analysis of GEMINI 1. Clin Exp Gastroenterol. 2020 Jun 11;13:211-220. doi: 10.2147/CEG.S248597. eCollection 2020. PMID 32606883
- [Derived] Dulai PS, Singh S, Vande Casteele N, Meserve J, Winters A, Chablaney S, Aniwan S, Shashi P, Kochhar G, Weiss A, Koliani-Pace JL, Gao Y, Boland BS, Chang JT, Faleck D, Hirten R, Ungaro R, Lukin D, Sultan K, Hudesman D, Chang S, Bohm M, Varma S, Fischer M, Shmidt E, Swaminath A, Gupta N, Rosario M, Jairath V, Guizzetti L, Feagan BG, Siegel CA, Shen B, Kane S, Loftus EV Jr, Sandborn WJ, Sands BE, Colombel JF, Lasch K, Cao C. Development and Validation of Clinical Scoring Tool to Predict Outcomes of Treatment With Vedolizumab in Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2020 Dec;18(13):2952-2961.e8. doi: 10.1016/j.cgh.2020.02.010. Epub 2020 Feb 13. PMID 32062041
- [Derived] Feagan BG, Schreiber S, Wolf DC, Axler JL, Kaviya A, James A, Curtis RI, Geransar P, Stallmach A, Ehehalt R, Bokemeyer B, Khalid JM, O'Byrne S. Sustained Clinical Remission With Vedolizumab in Patients With Moderate-to-Severe Ulcerative Colitis. Inflamm Bowel Dis. 2019 May 4;25(6):1028-1035. doi: 10.1093/ibd/izy323. PMID 30365009
- [Derived] Sandborn WJ, Colombel JF, Panaccione R, Dulai PS, Rosario M, Cao C, Barocas M, Lasch K. Deep Remission With Vedolizumab in Patients With Moderately to Severely Active Ulcerative Colitis: A GEMINI 1 post hoc Analysis. J Crohns Colitis. 2019 Feb 1;13(2):172-181. doi: 10.1093/ecco-jcc/jjy149. PMID 30285104
- [Derived] Feagan BG, Sandborn WJ, Colombel JF, Byrne SO, Khalid JM, Kempf C, Geransar P, Bhayat F, Rubin DT. Incidence of Arthritis/Arthralgia in Inflammatory Bowel Disease with Long-term Vedolizumab Treatment: Post Hoc Analyses of the GEMINI Trials. J Crohns Colitis. 2019 Jan 1;13(1):50-57. doi: 10.1093/ecco-jcc/jjy125. PMID 30203005
- [Derived] Feagan BG, Lasch K, Lissoos T, Cao C, Wojtowicz AM, Khalid JM, Colombel JF. Rapid Response to Vedolizumab Therapy in Biologic-Naive Patients With Inflammatory Bowel Diseases. Clin Gastroenterol Hepatol. 2019 Jan;17(1):130-138.e7. doi: 10.1016/j.cgh.2018.05.026. Epub 2018 May 29. PMID 29857145
- [Derived] Arijs I, De Hertogh G, Lemmens B, Van Lommel L, de Bruyn M, Vanhove W, Cleynen I, Machiels K, Ferrante M, Schuit F, Van Assche G, Rutgeerts P, Vermeire S. Effect of vedolizumab (anti-alpha4beta7-integrin) therapy on histological healing and mucosal gene expression in patients with UC. Gut. 2018 Jan;67(1):43-52. doi: 10.1136/gutjnl-2016-312293. Epub 2016 Oct 7. PMID 27802155
- [Derived] Feagan BG, Rubin DT, Danese S, Vermeire S, Abhyankar B, Sankoh S, James A, Smyth M. Efficacy of Vedolizumab Induction and Maintenance Therapy in Patients With Ulcerative Colitis, Regardless of Prior Exposure to Tumor Necrosis Factor Antagonists. Clin Gastroenterol Hepatol. 2017 Feb;15(2):229-239.e5. doi: 10.1016/j.cgh.2016.08.044. Epub 2016 Sep 14. PMID 27639327
- [Derived] Colombel JF, Sands BE, Rutgeerts P, Sandborn W, Danese S, D'Haens G, Panaccione R, Loftus EV Jr, Sankoh S, Fox I, Parikh A, Milch C, Abhyankar B, Feagan BG. The safety of vedolizumab for ulcerative colitis and Crohn's disease. Gut. 2017 May;66(5):839-851. doi: 10.1136/gutjnl-2015-311079. Epub 2016 Feb 18. PMID 26893500
- [Derived] Rosario M, Dirks NL, Gastonguay MR, Fasanmade AA, Wyant T, Parikh A, Sandborn WJ, Feagan BG, Reinisch W, Fox I. Population pharmacokinetics-pharmacodynamics of vedolizumab in patients with ulcerative colitis and Crohn's disease. Aliment Pharmacol Ther. 2015 Jul;42(2):188-202. doi: 10.1111/apt.13243. Epub 2015 May 20. PMID 25996351

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 211 investigative sites worldwide. The Induction Phase contained 2 cohorts. The eligibility criteria for both cohorts were identical. The purpose of Cohort 2 was to provide enough responders to power the Maintenance Phase primary efficacy analysis.
Pre-assignment Details: In Cohort 1, eligible patients who met entry criteria were randomized to treatment with double-blind vedolizumab 300 mg or placebo in a 3:2 ratio. All Cohort 2 patients were treated with open-label vedolizumab. In the Maintenance Phase participants were assigned to treatment groups based on their Induction Phase treatment and response to therapy.
Groups:
- Placebo: In the Induction Phase participants in Cohort 1 were randomized to receive double-blind placebo intravenous infusions at Week 0 and Week 2. Participants continued to receive placebo every 4 weeks from Week 6 through Week 50 during the Maintenance Phase, regardless of treatment response during induction.
- Induction Phase: DB Vedolizumab: In the Induction Phase participants in Cohort 1 were randomized to receive double-blind (DB) vedolizumab 300 mg, administered by intravenous infusion at Week 0 and Week 2.
- Induction Phase: OL Vedolizumab: In the Induction Phase participants in Cohort 2 received open-label (OL) vedolizumab 300 mg, administered by intravenous infusion at Week 0 and Week 2.
- Maintenance Phase: Placebo: Participants who received vedolizumab during the Induction Phase and demonstrated a clinical response at Week 6 were then randomized to receive double-blind treatment with placebo every 4 weeks up to Week 50 during the Maintenance Phase.
- Maintenance Phase: Vedolizumab Q8W: Participants who received vedolizumab during the Induction Phase and demonstrated a clinical response at Week 6 were then randomized to receive double-blind treatment with vedolizumab 300 mg every 8 weeks (Q8W) at Weeks 6, 14, 22, 30, 38, and 46, and, to maintain blinding, placebo infusions at Weeks 10, 18, 26, 34, 42, and 50.
- Maintenance Phase: Vedolizumab Q4W: Participants who received vedolizumab during the Induction Phase and demonstrated a clinical response at Week 6 were then randomized to receive double-blind treatment with vedolizumab 300 mg every 4 weeks (Q4W) from Week 6 to Week 50.
- Maintenance Phase: Non-responders: Participants who received vedolizumab during the Induction Phase who did not demonstrate a clinical response at Week 6 received open-label treatment with vedolizumab 300 mg every 4 weeks from Week 6 to Week 50.
Period: Induction Phase
Arm/Group | Placebo | Induction Phase: DB Vedolizumab | Induction Phase: OL Vedolizumab | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab Q8W | Maintenance Phase: Vedolizumab Q4W | Maintenance Phase: Non-responders
Started | 149 | 225 | 521 | 0 | 0 | 0 | 0
Completed | 135 | 218 | 485 | 0 | 0 | 0 | 0
Not Completed | 14 | 7 | 36 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 7 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 6 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 5 | 2 | 14 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 8 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0 | 0
Period: Maintenance Phase
Arm/Group | Placebo | Induction Phase: DB Vedolizumab | Induction Phase: OL Vedolizumab | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab Q8W | Maintenance Phase: Vedolizumab Q4W | Maintenance Phase: Non-responders
Started | 135 | 0 | 0 | 126 | 122 | 125 | 330
Completed | 30 | 0 | 0 | 48 | 77 | 84 | 135
Not Completed | 105 | 0 | 0 | 78 | 45 | 41 | 195
Not completed — Adverse Event | 12 | 0 | 0 | 15 | 7 | 6 | 16
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lack of Efficacy | 83 | 0 | 0 | 61 | 31 | 33 | 155
Not completed — Withdrawal by Subject | 6 | 0 | 0 | 2 | 5 | 2 | 20
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are provided for the Induction Phase Safety Population, defined as all participants, in both Cohort 1 and Cohort 2, who received any amount of study drug in the Induction Phase (Weeks 0-6), according to the actual study drug received.
Groups:
- Induction Phase: DB Vedolizumab: In the Induction Phase participants in Cohort 1 were randomized to receive double-blind vedolizumab 300 mg, administered by intravenous infusion at Week 0 and Week 2.
- Induction Phase: OL Vedolizumab: In the Induction Phase participants in Cohort 2 received open-label vedolizumab 300 mg, administered by intravenous infusion at Week 0 and Week 2.
- Total: Total of all reporting groups
Arm/Group | Placebo | Induction Phase: DB Vedolizumab | Induction Phase: OL Vedolizumab | Total
Number analyzed (Participants) | 149 | 225 | 521 | 895
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (12.50) | 40.1 (13.11) | 40.1 (13.27) | 40.3 (13.09)
Age, Customized [Number; unit: participants]
  < 35 | 53 | 86 | 214 | 353
  ≥ 35 | 96 | 139 | 307 | 542
Age, Customized [Number; unit: participants]
  < 65 | 142 | 217 | 503 | 862
  ≥ 65 | 7 | 8 | 18 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 93 | 220 | 370
  Male | 92 | 132 | 301 | 525
Race/Ethnicity, Customized [Number; unit: participants]
  White | 115 | 183 | 436 | 734
  Black | 2 | 5 | 5 | 12
  Asian | 32 | 36 | 67 | 135
  Other | 0 | 1 | 13 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 5 | 10 | 31 | 46
  Not Hispanic or Latino | 140 | 211 | 481 | 832
  Not reported | 4 | 4 | 9 | 17
Region of Enrollment [Number; unit: participants]
  Australia | 7 | 17 | 29 | 53
  Austria | 4 | 3 | 12 | 19
  Belgium | 7 | 14 | 35 | 56
  Bulgaria | 2 | 1 | 3 | 6
  Canada | 16 | 14 | 62 | 92
  Czech Republic | 7 | 12 | 19 | 38
  Denmark | 2 | 7 | 5 | 14
  Estonia | 1 | 4 | 5 | 10
  France | 1 | 3 | 13 | 17
  Germany | 0 | 1 | 16 | 17
  Greece | 0 | 1 | 4 | 5
  Hong Kong | 0 | 0 | 1 | 1
  Hungary | 2 | 6 | 8 | 16
  Iceland | 0 | 1 | 2 | 3
  India | 18 | 16 | 24 | 58
  Ireland | 0 | 0 | 1 | 1
  Israel | 0 | 1 | 1 | 2
  Italy | 1 | 9 | 11 | 21
  Korea, Republic of | 5 | 10 | 26 | 41
  Latvia | 1 | 2 | 0 | 3
  Malaysia | 5 | 2 | 2 | 9
  Netherlands | 1 | 0 | 2 | 3
  New Zealand | 0 | 5 | 6 | 11
  Norway | 2 | 1 | 6 | 9
  Poland | 2 | 6 | 52 | 60
  Russian Federation | 9 | 15 | 25 | 49
  Singapore | 0 | 0 | 1 | 1
  South Africa | 4 | 5 | 10 | 19
  Spain | 0 | 0 | 2 | 2
  Switzerland | 2 | 1 | 3 | 6
  Turkey | 0 | 3 | 3 | 6
  United Kingdom | 2 | 0 | 4 | 6
  United States | 47 | 64 | 127 | 238
Body Weight [Mean (Standard Deviation); unit: kg] — Body weight data only available for 148 participants in the placebo arm.
  kg | 72.4 (17.65) | 72.4 (17.11) | 74.2 (19.32) | 73.4 (18.51)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI data only available for 148 participants in the placebo arm.
  kg/m^2 | 24.6 (5.11) | 24.9 (4.85) | 25.3 (6.05) | 25.1 (5.62)
Duration of Ulcerative Colitis [Mean (Standard Deviation); unit: years] — Duration of ulcerative colitis data only available for 519 participants in the Induction Phase: OL Vedolizumab arm.
  years | 7.1 (7.25) | 6.1 (5.08) | 7.2 (6.61) | 6.9 (6.39)
Categorical Duration of Ulcerative Colitis [Number; unit: participants]
  < 1 year | 13 | 13 | 38 | 64
  ≥1 - < 3 years | 44 | 63 | 121 | 228
  ≥ 3 - < 7 years | 39 | 77 | 163 | 279
  ≥ 7 years | 53 | 72 | 197 | 322
  Missing | 0 | 0 | 2 | 2
Baseline Mayo Score [Mean (Standard Deviation); unit: units on a scale] — The Mayo Score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 components: two that are patient reported (rectal bleeding and stool frequency), a global assessment by the physician, and an endoscopic subscore. Each component is scored on a scale from 0 to 3 and the complete score ranges from 1 to 12 (higher scores indicate greater disease activity).
  units on a scale | 8.6 (1.68) | 8.5 (1.78) | 8.6 (1.76) | 8.6 (1.75)
Baseline Disease Activity [Number; unit: participants]
  Complete Mayo score < 6 | 5 | 6 | 14 | 25
  Complete Mayo score of 6 to 8 (inclusive) | 70 | 105 | 249 | 424
  Complete Mayo score of 9 to 12 (inclusive) | 74 | 114 | 258 | 446
Baseline Fecal Calprotectin [Mean (Standard Deviation); unit: μg/g] — Number of participants for whom baseline fecal calprotectin data were available were 139, 213, and 505, respectively.
  μg/g | 2369.9 (3258.82) | 2552.2 (3800.36) | 1442.7 (1855.61) | 1868.8 (2753.28)
Categorical Baseline Fecal Calprotectin [Number; unit: participants]
  ≤ 250 μg/g | 27 | 37 | 94 | 158
  > 250 to ≤ 500 μg/g | 20 | 20 | 82 | 122
  > 500 μg/g | 92 | 156 | 329 | 577
  Missing | 10 | 12 | 16 | 38
Disease Localization [Number; unit: participants]
  Proctosigmoiditis | 22 | 25 | 69 | 116
  Left-sided colitis | 59 | 92 | 188 | 339
  Extensive colitis | 18 | 25 | 66 | 109
  Pancolitis | 50 | 83 | 198 | 331
Smoking Status [Number; unit: participants]
  Current smoker | 11 | 12 | 32 | 55
  Nonsmoker | 88 | 145 | 322 | 555
  Former smoker | 50 | 68 | 167 | 285
History of Extraintestinal Manifestations [Number; unit: participants]
  Yes | 44 | 74 | 180 | 298
  No | 105 | 151 | 341 | 597

OUTCOME MEASURES:

1. Primary Outcome: Induction Phase: Percentage of Participants With a Clinical Response at Week 6
Description: Clinical response is defined as a reduction in complete Mayo score of ≥ 3 points and ≥ 30% from Baseline with an accompanying decrease in rectal bleeding subscore of ≥ 1 point or absolute rectal bleeding subscore of ≤ 1 point.
  The Mayo Score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 components: two that are patient reported (rectal bleeding and stool frequency), a global assessment by the physician, and an endoscopic subscore. Each component is scored on a scale from 0 to 3 and the complete score ranges from 1 to 12 (higher scores indicate greater disease activity).
  All participants who prematurely discontinued for any reason were considered as not achieving clinical response.
Time Frame: Baseline and Week 6
Population: Induction Study Intent-to-treat (ITT) population which consisted of all randomized patients in Cohort 1 who received any amount of blinded study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Participants in Cohort 1 received double-blind placebo intravenous infusions at Week 0 and Week 2 in the Induction Phase.
- DB Vedolizumab: Participants in Cohort 1 received double-blind vedolizumab 300 mg, administered by intravenous infusion at Week 0 and Week 2 in the Induction Phase.
Arm/Group | Placebo | DB Vedolizumab
Number analyzed (Participants) | 149 | 225
percentage of participants | 25.5 [18.5 to 32.5] | 47.1 [40.6 to 53.6]
Statistical Analysis 1: Comparison: Placebo vs DB Vedolizumab; The primary comparison of the Induction Phase was tested using the Cochran-Mantel-Haenszel (CMH) chi-square test at a 5% significance level, with stratification according to the stratification factors (concomitant use of oral corticosteroids and previous exposure to tumor necrosis factor alpha (TNFα) antagonists or concomitant immunomodulator [6-mercaptopurine or azathioprine] use); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 21.7, 95% CI 2-sided [11.6 to 31.7]

2. Primary Outcome: Maintenance Phase: Percentage of Participants in Clinical Remission at Week 52
Description: Clinical Remission is defined as a complete Mayo score of ≤ 2 points and no individual subscore > 1 point.
  The Mayo Score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 components: two that are patient reported (rectal bleeding and stool frequency), a global assessment by the physician, and an endoscopic subscore. Each component is scored on a scale from 0 to 3 and the complete score ranges from 1 to 12 (higher scores indicate greater disease activity).
  All participants who prematurely discontinued for any reason were considered as not achieving clinical remission.
Time Frame: Week 52
Population: Maintenance Study ITT Population, defined as all randomized participants who received vedolizumab during the Induction Phase and met the protocol definition of clinical response at Week 6, as assessed by the investigator, were randomized, and received any amount of double-blind study drug in the Maintenance Phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Participants who received vedolizumab during the Induction Phase and demonstrated a clinical response at Week 6 were randomized to receive double-blind treatment with placebo every 4 weeks up to Week 50 during the Maintenance Phase.
- Vedolizumab Q8W: Participants who received vedolizumab during the Induction Phase and demonstrated a clinical response at Week 6 were randomized to receive double-blind treatment with vedolizumab 300 mg every 8 weeks (Q8W) from Week 6 to Week 50.
- Vedolizumab Q4W: Participants who received vedolizumab during the Induction Phase and demonstrated a clinical response at Week 6 were randomized to receive double-blind treatment with vedolizumab 300 mg every 4 weeks (Q4W) from Week 6 to Week 50.
Arm/Group | Placebo | Vedolizumab Q8W | Vedolizumab Q4W
Number analyzed (Participants) | 126 | 122 | 125
percentage of participants | 15.9 [9.5 to 22.3] | 41.8 [33.1 to 50.6] | 44.8 [36.1 to 53.5]
Statistical Analysis 1: Comparison: Placebo vs Vedolizumab Q8W; The Hochberg method was applied to control the overall Type I error rate at a 5% significance level. If both P-values were ≤ 0.05, both dose regimens were to be declared significant. If 1 of the P-values for the 2 dose comparisons was > 0.05, the other P-value was to be tested at the 0.025 level and declared significant only if the P-value was ≤ 0.025. If neither dose was declared significant for the primary endpoint, no further testing was to be conducted; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — P-value is based on the CMH chi-square test, with 3 stratification factors: concomitant use of oral corticosteroids; previous exposure to TNFα antagonists or concomitant immunomodulator use; enrollment in Cohort 1 or 2 in the Induction Phase; Risk Difference (RD) = 26.1, 95% CI 2-sided [14.9 to 37.2]
Statistical Analysis 2: Comparison: Placebo vs Vedolizumab Q4W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 29.1, 95% CI 2-sided [17.9 to 40.4]

3. Secondary Outcome: Induction Phase: Percentage of Participants in Clinical Remission at Week 6
Description: as for outcome 2
Time Frame: Week 6
Population: Induction Study ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | DB Vedolizumab
Number analyzed (Participants) | 149 | 225
percentage of participants | 5.4 [1.7 to 9.0] | 16.9 [12.0 to 21.8]
Statistical Analysis 1: Comparison: Placebo vs DB Vedolizumab; To maintain the overall Type I error rate at 5%, the key secondary assessments were performed sequentially (closed sequential method). The first secondary endpoint was to be tested only if the primary comparison was significant and the second key secondary endpoint was to be tested only if the first secondary endpoint was significant for vedolizumab; Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel — P-value is based on the CMH chi-square test, with stratification according to: 1) concomitant use of oral corticosteroids (yes/no); and 2) previous exposure to TNFα antagonists or concomitant immunomodulator use (yes/no); Risk Difference (RD) = 11.5, 95% CI 2-sided [4.7 to 18.3]

4. Secondary Outcome: Induction Phase: Percentage of Participants With Mucosal Healing at Week 6
Description: Mucosal healing is defined as a Mayo endoscopic subscore of ≤ 1 point.
  The Mayo Score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 components: two that are patient reported (rectal bleeding and stool frequency), a global assessment by the physician, and an endoscopic subscore. Endoscopic findings were scored on a scale from 0 to 3 as follows:
  0 = Normal or inactive disease; 1 = Mild disease (erythema, decreased vascular pattern, mild friability); 2 = Moderate disease (marked erythema, lack of vascular pattern, friability, erosions); 3 = Severe disease (spontaneous bleeding, ulceration).
  All participants who prematurely discontinued for any reason were considered as not achieving mucosal healing.
Time Frame: Week 6
Population: Induction Study ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | DB Vedolizumab
Number analyzed (Participants) | 149 | 225
percentage of participants | 24.8 [17.9 to 31.8] | 40.9 [34.5 to 47.3]
Statistical Analysis 1: Comparison: Placebo vs DB Vedolizumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0012, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Risk Difference (RD) = 16.1, 95% CI [6.4 to 25.9]

5. Secondary Outcome: Maintenance Phase: Percentage of Participants With Durable Clinical Response
Description: Durable clinical response is defined as reduction in complete Mayo score of ≥ 3 points and ≥ 30% from Baseline (Week 0) with an accompanying decrease in rectal bleeding subscore of ≥ 1 point or absolute rectal bleeding subscore of ≤ 1 point at both Weeks 6 and 52. The Mayo Score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 components: two that are patient reported (rectal bleeding and stool frequency), a global assessment by the physician, and an endoscopic subscore. Each component is scored on a scale from 0 to 3 and the complete score ranges from 1 to 12 (higher scores indicate greater disease activity).
  All participants who prematurely discontinued for any reason were considered as not achieving durable clinical response.
Time Frame: Baseline, Week 6 and Week 52
Population: Maintenance Study ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Vedolizumab Q8W | Vedolizumab Q4W
Number analyzed (Participants) | 126 | 122 | 125
percentage of participants | 23.8 [16.4 to 31.2] | 56.6 [47.8 to 65.4] | 52.0 [43.2 to 60.8]
Statistical Analysis 1: Comparison: Placebo vs Vedolizumab Q8W; To maintain the overall Type I error rate at 5% for the 2 dose regimen comparisons for each key secondary endpoint, the Hochberg method was used as described for the primary outcome measure. To further maintain the overall Type I error rate at 5%, the key secondary endpoints were also performed sequentially. The first was tested only if 1 or both of the primary comparisons were significant and the next endpoint was tested only if the previous endpoint was significant for at least 1 dose; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 32.8, 95% CI 2-sided [20.8 to 44.7]
Statistical Analysis 2: Comparison: Placebo vs Vedolizumab Q4W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 28.5, 95% CI 2-sided [16.7 to 40.3]

6. Secondary Outcome: Maintenance Phase: Percentage of Participants With Mucosal Healing at Week 52
Description: as for outcome 4
Time Frame: Week 52
Population: Maintenance Study ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Vedolizumab Q8W | Vedolizumab Q4W
Number analyzed (Participants) | 126 | 122 | 125
percentage of participants | 19.8 [12.9 to 26.8] | 51.6 [42.8 to 60.5] | 56.0 [47.3 to 64.7]
Statistical Analysis 1: Comparison: Placebo vs Vedolizumab Q8W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 32.0, 95% CI 2-sided [20.3 to 43.8]
Statistical Analysis 2: Comparison: Placebo vs Vedolizumab Q4W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 36.3, 95% CI 2-sided [24.4 to 48.3]

7. Secondary Outcome: Maintenance Phase: Percentage of Participants With Durable Clinical Remission
Description: Durable clinical remission is defined as complete Mayo score of ≤ 2 points and no individual subscore > 1 point at both Weeks 6 and 52. The Mayo Score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 components: two that are patient reported (rectal bleeding and stool frequency), a global assessment by the physician, and an endoscopic subscore. Each component is scored on a scale from 0 to 3 and the complete score ranges from 1 to 12 (higher scores indicate greater disease activity).
  All participants who prematurely discontinued for any reason were considered as not achieving durable clinical remission.
Time Frame: Week 6 and Week 52
Population: Maintenance Study ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Vedolizumab Q8W | Vedolizumab Q4W
Number analyzed (Participants) | 126 | 122 | 125
percentage of participants | 8.7 [3.8 to 13.7] | 20.5 [13.3 to 27.7] | 24.0 [16.5 to 31.5]
Statistical Analysis 1: Comparison: Placebo vs Vedolizumab Q8W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0079, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 11.8, 95% CI 2-sided [3.1 to 20.5]
Statistical Analysis 2: Comparison: Placebo vs Vedolizumab Q4W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 15.3, 95% CI 2-sided [6.2 to 24.4]

8. Secondary Outcome: Maintenance Phase: Percentage of Participants With Corticosteroid-free Remission at Week 52
Description: Clinical Remission is defined as a complete Mayo score of ≤ 2 points and no individual subscore > 1 point. Corticosteroid-free clinical remission is defined as participants using oral corticosteroids at baseline (Week 0) who discontinued corticosteroids and were in clinical remission at Week 52.
  The Mayo Score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 components: two that are patient reported (rectal bleeding and stool frequency), a global assessment by the physician, and an endoscopic subscore. Each component is scored on a scale from 0 to 3 and the complete score ranges from 1 to 12 (higher scores indicate greater disease activity).
  All participants who prematurely discontinued for any reason were considered as not achieving corticosteroid-free remission.
Time Frame: Week 52
Population: Maintenance Study ITT Population, participants who were on corticosteroids at Baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Vedolizumab Q8W | Vedolizumab Q4W
Number analyzed (Participants) | 72 | 70 | 73
percentage of participants | 13.9 [5.9 to 21.9] | 31.4 [20.6 to 42.3] | 45.2 [33.8 to 56.6]
Statistical Analysis 1: Comparison: Placebo vs Vedolizumab Q8W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0120, Cochran-Mantel-Haenszel — P-value based on the CMH chi-square test, with 3 stratification factors: concomitant use of oral corticosteroids; previous exposure to TNFα antagonists or concomitant immunomodulator use; enrollment in Cohort 1 or 2 in the Induction Phase; Risk Difference (RD) = 17.6, 95% CI 2-sided [3.9 to 31.3]
Statistical Analysis 2: Comparison: Placebo vs Vedolizumab Q4W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 31.4, 95% CI 2-sided [16.6 to 46.2]

ADVERSE EVENTS:
Time Frame: From the start of the Induction Phase until a final on-study safety assessment at Week 66 (or Final Safety visit 16 weeks after the last dose).
Groups:
- Placebo: Participants who received double-blind placebo intravenous infusions in the Induction Phase and continued to receive placebo during the Maintenance Phase.
- Vedolizumab Then Placebo: Participants who received vedolizumab during the Induction Phase and were then randomized to receive placebo during the Maintenance Phase.
- Vedolizumab: Participants who received vedolizumab during the Induction Phase and continued to receive vedolizumab during the Maintenance Phase. This includes participants who had a clinical response at Week 6 and were randomized to vedolizumab every 4 weeks or every 8 weeks in the Maintenance Phase, participants who did not achieve a clinical response at Week 6 and continued to receive vedolizumab every 4 weeks for the duration of the study, and participants who withdrew during the Induction phase.
Arm/Group | Placebo | Vedolizumab Then Placebo | Vedolizumab
Serious Adverse Events (participants affected / at risk) | 17/149 | 20/126 | 77/620
Other Adverse Events (participants affected / at risk) | 67/149 | 69/126 | 321/620
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=149) | Vedolizumab Then Placebo (N=126) | Vedolizumab (N=620)
Colitis ulcerative (Gastrointestinal disorders) | 10 | 7 | 47
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Colon dysplasia (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 2
Wound infection (Infections and infestations) | 0 | 0 | 2
Perirectal abscess (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Cholangitis suppurative (Infections and infestations) | 0 | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Pulpitis dental (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 2 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 0 | 0
Pericoronitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Accidental poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis sclerosing (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Haemoglobin decrease (Investigations) | 0 | 1 | 1
Lipase increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Arteriosclerosis obliterans (Vascular disorders) | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Sarcoidosis (Immune system disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=149) | Vedolizumab Then Placebo (N=126) | Vedolizumab (N=620)
Nasopharyngitis (Infections and infestations) | 11 | 15 | 80
Upper respiratory tract infection (Infections and infestations) | 8 | 13 | 52
Bronchitis (Infections and infestations) | 5 | 7 | 23
Colitis ulcerative (Gastrointestinal disorders) | 20 | 22 | 57
Nausea (Gastrointestinal disorders) | 11 | 8 | 38
Abdominal pain (Gastrointestinal disorders) | 7 | 2 | 34
Headache (Nervous system disorders) | 13 | 15 | 80
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 15 | 56
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 36
Anaemia (Blood and lymphatic system disorders) | 10 | 4 | 35
Fatigue (General disorders) | 5 | 5 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.